CLINICAL TRIAL: NCT00913770
Title: Models of Screening, Brief Intervention With a Facilitated Referral to Treatment (SBIRT) for Opioid Patients in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0808004132; 1R01DA025991-01 (NIH)
Record Dates: First submitted 2009-06-01; First posted 2009-06-04 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Opiate Addiction
Keywords: opioid dependence; buprenorphine; brief intervention
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- SC (No Intervention): Standard Care
- SBIRT (Experimental): Screening, Brief Intervention and Facilitated Referral to Treatment
  Interventions: Behavioral: Brief Negotiation Interview (BNI)
- SBI+Bup (Experimental): Screening, Brief Intervention and Buprenorphine initiation
  Interventions: Behavioral: Brief Negotiation Interview (BNI); Drug: Buprenorphine Initiation

INTERVENTIONS:
Behavioral: Brief Negotiation Interview (BNI) — Brief Negotiation Interview (BNI) is a manual-guided therapy that is designed to be feasible in the ED setting. The purpose of the BNI is to assist patients in recognizing and changing their drug use and HIV risk behaviors. It combines techniques based on motivational interviewing and a stage-model of change. The main goal of the interview is to decrease the subject's ambivalence about signing up for a formal drug treatment program.
  Arms: SBI+Bup; SBIRT
Drug: Buprenorphine Initiation
  Arms: SBI+Bup

SUMMARY:
Patients with heroin and prescription opioid dependence are at increased risk for adverse health consequences and often utilize the Emergency Department (ED) as their source of medical care. Screening, brief intervention and referral to treatment has been effective in decreasing high risk behaviors such as alcohol and tobacco use, and unsafe sexual practices. The data on the effectiveness of brief interventions with opioid dependence is limited. This prospective, randomized controlled trial of opioid dependent subjects (N=360) will compare two models of brief intervention with a control condition. ED patients with opioid dependence will be randomized to either: (1)Screening, Brief Intervention with a Facilitated Referral to Treatment (SBIRT); (2) Screening, Brief Intervention with ED initiated Buprenorphine Treatment (SBI+Bup); or (3) standard care (SC) which includes a handout detailing substance abuse treatment centers in the area. The primary outcome will be self-reported engagement in formal substance abuse treatment at 30 days, verified by contact with the treatment program. Other outcomes measured at 30 days, 2, 6 and 12 months include changes in opioid use (self-report and urine toxicology analysis), HIV risk behaviors, and health care service utilization. The three interventions will also be compared on their cost-effectiveness. We will test the hypotheses that SBI+Bup will be superior to SBIRT and SC, and SBIRT will be superior to SC in (1)increasing the proportion of patients engaged in formal substance abuse treatment at 30 days; (2) reducing illicit opioid use; (3) reducing HIV risk behaviors; and (4) reducing health care service utilization. In addition, we hypothesize that the societal costs of SBI+Bup, per number of days of opioid abstinence, will be cost effective relative to SBIRT or SC; and that SBIRT will be cost effective relative to SC. Data analyses will be conducted on the intention to treat sample of randomized patients. This study, conducted by a research team with extensive experience evaluating brief interventions and treatments for opioid dependence, will be unique in its: (1) comparison of two models of brief intervention with standard care; (2) inclusion of an ED initiated treatment arm; (3) use of manual-guided interventions with systematic assessment of adherence and competence; and (4)collection of detailed cost data to help guide future healthcare policy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the adult ED at Yale-New Haven Hospital (YNHH) who are:

  1. 18 years or older,
  2. meet criteria for opioid dependence as measured by the Mini-SCID, and
  3. have a positive urine toxicology for opiates.

Exclusion Criteria:

* Inability to read or understand English
* Currently receiving formal substance abuse treatment
* Current suicide or homicidal risk
* Current psychotic disorder
* Life-threatening or unstable medical or psychiatric condition requiring hospital admission
* Unable to provide 2 phone contact numbers
* Unwilling to be randomized and/or follow up as per study protocol, including release of information to assess treatment engagement at 30-days
* Requiring opioid agonist medication for a pain-related diagnosis (contraindication to buprenorphine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2008-09; Primary Completion 2013-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail D'Onofrio, MD, MS, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut

REFERENCES:
- [Result] D'Onofrio G, O'Connor PG, Pantalon MV, Chawarski MC, Busch SH, Owens PH, Bernstein SL, Fiellin DA. Emergency department-initiated buprenorphine/naloxone treatment for opioid dependence: a randomized clinical trial. JAMA. 2015 Apr 28;313(16):1636-44. doi: 10.1001/jama.2015.3474. PMID 25919527
- [Result] Busch SH, Fiellin DA, Chawarski MC, Owens PH, Pantalon MV, Hawk K, Bernstein SL, O'Connor PG, D'Onofrio G. Cost-effectiveness of emergency department-initiated treatment for opioid dependence. Addiction. 2017 Nov;112(11):2002-2010. doi: 10.1111/add.13900. Epub 2017 Aug 16. PMID 28815789
- [Result] D'Onofrio G, Chawarski MC, O'Connor PG, Pantalon MV, Busch SH, Owens PH, Hawk K, Bernstein SL, Fiellin DA. Emergency Department-Initiated Buprenorphine for Opioid Dependence with Continuation in Primary Care: Outcomes During and After Intervention. J Gen Intern Med. 2017 Jun;32(6):660-666. doi: 10.1007/s11606-017-3993-2. Epub 2017 Feb 13. PMID 28194688
- [Derived] Nielsen S, Tse WC, Larance B. Opioid agonist treatment for people who are dependent on pharmaceutical opioids. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD011117. doi: 10.1002/14651858.CD011117.pub3. PMID 36063082

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care: Standard Care including receiving a referral.
- SBIRT: Screening, Brief Intervention and Facilitated Referral to Treatment
  Brief Intervention: Brief Negotiated Intervention (BNI) is a manual-guided therapy that is designed to be feasible in the ED setting. The purpose of the BNI is to assist patients in recognizing and changing their drug use and HIV risk behaviors. It combines techniques based on motivational interviewing and a stage-model of change. The main goal of the interview is to decrease the subject's ambivalence about signing up for a formal drug treatment program.
- SBI+Bup: Screening, Brief Intervention and Buprenorphine initiation
  Brief Intervention with Buprenorphine initiation: Brief Negotiated Intervention is a manual-guided therapy designed for ED setting. Purpose- to assist patients recognize/change drug use and HIV risks. It combines techniques based on motivational interviewing and a stage-model of change. Goal- to decrease subject's ambivalence about accepting ED initiated buprenorphine treatment. Patients inducted onto buprenorphine in ED or home, based on level of withdrawal. ED induction goal- 8 mg first day. Home induction goal- 8 mg first day. Subjects receive supportive counseling and education by trained nurses in the PCC (seen within 24-72 hours of their ED visit). Following an initial 45-minute evaluation, the physician will administer Primary Care Management (PCM) weekly for 2 weeks, then every 2 weeks for 4 weeks and then monthly.
Period: Overall Study
Arm/Group | Standard Care | SBIRT | SBI+Bup
Started | 104 | 111 | 114
Completed | 69 | 82 | 93
Not Completed | 35 | 29 | 21
Not completed — Unable to contact | 24 | 19 | 13
Not completed — Refused | 11 | 10 | 8

BASELINE CHARACTERISTICS:
Population: Baseline population description is the number of subjects randomized to study arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | SBIRT | SBI+Bup | Total
Number analyzed (Participants) | 104 | 111 | 114 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (10.6) | 31.9 (9.7) | 31 (9.8) | 31.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 28 | 78
  Male | 81 | 84 | 86 | 251

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Engagement in Formal Substance Abuse Treatment at 30 Days (Verified by Contact With the Treatment Program)
Description: Defined as enrollment and receiving formal addiction treatment on the 30th day following randomization. This is assessed by direct contact with facility, clinician, or both.
Time Frame: 30 days post randomization
Population: All subjects who were randomized to receive treatment were included in the primary analysis. 2 subjects were lost to follow up in the standard of care arm which is why 102 are included in the analysis instead of 104
Measure: Mean (95% Confidence Interval); unit: Mean Number of Outpatient Visits
Arm/Group | Standard Care | SBIRT | SBI+Bup
Number analyzed (Participants) | 102 | 111 | 114
Mean Number of Outpatient Visits | 4.99 [3.1 to 6.8] | 5.67 [4.0 to 7.4] | 3.71 [2.1 to 5.3]

2. Secondary Outcome: Days of Self-reported Illicit Opioid Use in the Past 7 Days
Time Frame: 30 days post randomization
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Mean Number of Days
Arm/Group | Standard Care | SBIRT | SBI+Bup
Number analyzed (Participants) | 102 | 111 | 114
Mean Number of Days | 2.3 [1.7 to 3.0] | 2.4 [1.8 to 3.0] | 0.9 [0.5 to 1.3]

ADVERSE EVENTS:
Arm/Group | Standard Care | SBIRT | SBI+Bup
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/111 | 0/114
Other Adverse Events (participants affected / at risk) | 0/104 | 0/111 | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes